CLINICAL TRIAL: NCT05319743
Title: Evaluating the Quality and Value of U.S. Ambulatory Care Delivered Among Medicaid Expansion States and Non-Expansion States, 2012-2015
Brief Title: Evaluating Quality and Value of US Ambulatory Care Delivered Among Medicaid Expansion/Non-Expansion States, 2012-2015
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, John N. Mafi, MD, MPH, Associate Professor of Medicine, University of California, Los Angeles
Other Study IDs: 22-001139
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Medicaid Expansion
Keywords: High-value care; Low-value care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medicaid expansion states: Eight Medicaid expansion states: (experimental group): Arizona, California, Illinois, Massachusetts, New Jersey, Ohio, Washington
  Interventions: Other: Medicaid Expansion
- Non-Medicaid expansion states: Five states that did not expand Medicaid (control group): Florida, Georgia, North Carolina, Texas, Virginia

INTERVENTIONS:
Other: Medicaid Expansion — Expansion of Medicaid, 01/01/2014
  Groups: Medicaid expansion states

SUMMARY:
Quasi-experimental pre-post analysis of the rate of high-value and low-value care services between states that expanded Medicaid and states that did not expand Medicaid January 1, 2014, for adult ambulatory visits, using visit-level survey data from the National Ambulatory Medical Care Survey January 1, 2012 - December 31, 2015.

DETAILED DESCRIPTION:
Data Source: Visit level data obtained from the National Ambulatory Medical Care Survey (NAMCS) between January 1, 2012-December 31, 2015.

Identification of Observations (Visits) for Primary Analysis: Adult visits in states that did expand Medicaid January 1, 2014 (experimental group) and states that did not expand Medicaid January 1, 2014 (control group). Eight Medicaid expansion states (experimental group): Arizona, California, Illinois, Massachusetts, New Jersey, Ohio, Washington Five states that did not expand Medicaid (control group): Florida, Georgia, North Carolina, Texas, Virginia. Visits will be included only if they could receive a low value service (visits for back pain, headache, general medical exam, URI) or high value service (visits with patients who have CAD, DM, CVD, Depression, CHF, Osteoporosis and no exclusion to receive the indicated high value service) when evaluating low value service counts and high value service counts respectively as opposed to all adult visits regardless of the opportunity to receive a high value or low value care service (e.g. visit for hand pain and none of the high or low value areas above.)

Identification of Observations (Visits) for Secondary Analyses: Medicaid patient subpopulation will be defined as those visits for primary analysis that are coded with Medicaid as a pay type for the visit. "New" Medicaid patient subpopulation will be defined as those visits for primary analysis that are coded with Medicaid as a pay type, have not seen before, to a provider who is accepting new patients and accepts Medicaid for new patients.

Create Indicator Variables for Primary and Secondary Outcome Analyses: Develop a set of low value and high value services with distinct inclusion and exclusion criteria for each service. Create indicator variable for each high value and low value service. Low value care measures (Imaging for Low Back Pain, Opioid for Low Back Pain, Opioid for Headache, Imaging for Headache, Antibiotic for Upper Respiratory Infection, General Medical Examination with ECG ordered, General Medical Examination with Urinalysis ordered.) High value care measures (Antiplatelet for CAD, Beta Blocker for CAD, Statin for CAD, Anticoagulation for Atrial Fibrillation, Statin for DM, Antiplatelet CVD, Treatment for Depression, Beta Blocker for CHF, ACE/ARB/ARNI for CHF, Treatment for Osteoporosis)

Analysis: Evaluate for pre-intervention (Medicaid Expansion) parallel trends (This has already been established). Then perform pre-post difference-in-differences analyses of primary and secondary outcomes between the experimental group (states that expanded Medicaid) and control group (states that did not expand Medicaid). Regression analysis will be performed to adjust for respondent age, sex, race/ethnicity, number of chronic illnesses, and clinic rural/urban location. Stratified models based on payer type will allow for analyses of the Medicaid population. Perform sensitivity analyses of primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Visits between 01/01/2012 and 12/31/2015

Exclusion Criteria:

* <18 years old
* Visits before 01/01/2012
* Visits after 12/31/2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NAMCS Adult Visits between 01/01/2012 and 12/31/2015. The data source is a nationally representative probability sample of U.S. ambulatory care visits
Sampling Method: Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of low-value and high-value services for adult ambulatory visits. | pre (01/01/2012 - 12/31/2013) and post (01/01/2014 - 12/31/2015) Medicaid expansion
  Ex. Numerator = count of high value services provided for adult visits in Medicaid expansion states in 2012/ Denominator = Count of adult visits in Medicaid expansion state in 2012 that had the potential to receive a high value service.

SECONDARY OUTCOMES:
Adult ambulatory visit volume changes | pre (01/01/2012 - 12/31/2013) and post (01/01/2014 - 12/31/2015) Medicaid expansion
  All adults, Medicaid adults, "New" Medicaid adults
Rate of low-value and high-value services for Medicaid adult ambulatory visits | pre (01/01/2012 - 12/31/2013) and post (01/01/2014 - 12/31/2015) Medicaid expansion
  Ex. Numerator = count of high value services provided for Medicaid adult visits in Medicaid expansion states in 2012/ Denominator = Count of Medicaid adult visits in Medicaid expansion state in 2012 that had the potential to receive a high value service
Rate of low-value and high-value services for "New" Medicaid adult ambulatory visits. | pre (01/01/2012 - 12/31/2013) and post (01/01/2014 - 12/31/2015) Medicaid expansion
  Ex. Numerator = count of high value services provided for "New" Medicaid adult visits in Medicaid expansion states in 2012/ Denominator = Count of "New" Medicaid adult visits in Medicaid expansion state in 2012 that had the potential to receive a high value service.

OTHER OUTCOMES:
Sensitivity analysis: repeat primary and secondary analysis with all adult visits, Medicaid visits, and "New" Medicaid visits | pre (01/01/2012 - 12/31/2013) and post (01/01/2014 - 12/31/2015) Medicaid expansion
  1. Repeat primary and secondary analysis with all adult visits, Medicaid visits and "New" Medicaid visits with a denominator of all visits (not the denominator of visits with potential to receive low or high value service as described for the primary analyses)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publicly available NAMCS data